CLINICAL TRIAL: NCT03594734
Title: Efficacy of an Evidence-based Weight-loss Intervention Post Traumatic Brain Injury
Brief Title: Group Lifestyle Balance™ for Individuals With Traumatic Brain Injury (GLB-TBI)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency); University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: BSWRI 017-482
Record Dates: First submitted 2018-06-28; First posted 2018-07-20 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic Brain Injury; Group Lifestyle Balance; Weight-Loss
MeSH Terms: conditions — Brain Injuries, Traumatic; Weight Loss

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial (RCT).
  Participants will be randomized into two group: (1) the GLB Intervention Group and (2) the Attention Control Group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GLB Weight-Loss Intervention (Experimental): The GLB program, adapted for individuals with TBI, will be delivered to participants over a 12-month period, divided into 22 in-person or virtual, group sessions. The intervention promotes 5-7% weight-loss by reducing calories and increasing exercise (150 minutes of moderate physical activity per week).
  Interventions: Behavioral: Group Lifestyle Balance™
- Attention Control Group (Active Comparator): The attention control group will meet at the same frequency as the GLB-TBI group over a 12-month period. The attention control group will receive education composed of the content from the TBI Model Systems Knowledge Translation Center's factsheets. No education on weight-loss strategies will be provided.
  Interventions: Other: Attention Control Group

INTERVENTIONS:
Behavioral: Group Lifestyle Balance™ — The Group Lifestyle Balance™ (GLB) program is a self-management intervention that has been shown to result in weight-loss and reduce the risk for Type 2 diabetes through increased physical activity and healthy eating behaviors in the general population. The GLB program curriculum used in this RCT will be adapted for individuals with TBI.
  Arms: GLB Weight-Loss Intervention
Other: Attention Control Group — The attention control group will receive the same contact or "attention" as the intervention group. The attention control group will meet at the same frequency as the intervention group. Education for the sessions will be composed of content from the TBI Model Systems Knowledge Translation Center's factsheets. General topics will include discussion on (1) healthy brain and effects of TBI on cognitive, emotional, and behavioral functioning, (2) expectations for recovery, (3) preventative and management strategies for common TBI sequela (e.g. inability and impulsivity), (4) stress management, (5), signs and symptoms of depression, and (6) strategies for effective communication.
  Arms: Attention Control Group

SUMMARY:
The purpose of this RCT is to examine the efficacy of a Group Lifestyle Balance™ (GLB) program adapted for people with traumatic brain injury (TBI) on primary (weight) and secondary outcomes at 3, 6, 12, and 18 months from enrollment into the program.

DETAILED DESCRIPTION:
Weight gain is common among people with TBI. Weight gain greatly increases the risk of chronic diseases such as diabetes, metabolic syndrome, pulmonary and heart disease. Approaches to weight-loss are lacking, yet necessary, due to the unique physiological and cognitive needs of persons with TBI. There is evidence that interventions that improve physical activity and healthy eating behaviors concurrently offer greatest potential for weight-loss. The Group Lifestyle Balance™ (GLB) intervention is a 12-month, evidence-based weight-loss program that has been used extensively with the general population, but not with people with TBI. The investigators modified the program to meet the needs of people with a TBI (GLB-TBI) and a pilot study with 20 individuals with TBI demonstrated that participation resulted in 5% weight-loss (10.2±13lbs) warranting a rigorous RCT. In addition, the investigators propose to integrate a mobile app into the GLB-TBI as 94% of pilot participants indicated that text messaging to support weight-loss would have been "very helpful" to boost motivation.

The proposed study consists of four specific aims.

Specific Aim 1: To examine the efficacy of the GLB-TBI compared to an attention control at 3, 6, 12, and 18 months from baseline using a randomized controlled trial.

Specific Aim 2: To examine participant compliance to GLB-TBI intervention components and its association with their outcomes:

Aim 2.1: To determine participant compliance with specific components of the GLB-TBI, including: (1) session attendance (2) self-monitoring of dietary and activity behaviors and (3) activity tracking of step count through accelerometer data.

Aim 2.2: To determine if compliance with the GLB-TBI is associated with improvement in primary (weight) and secondary outcomes (step count; waist circumference; blood pressure; HbA1c and lipid panel; functional measures; and quality of life).

Specific Aim 3: To assess feasibility (compliance, usability) of adding a smartphone application at week 12 of the GLB-TBI program and attention control condition to enhance participant engagement.

Specific Aim 4: Ascertain maintenance of primary (weight) and additional secondary outcomes (step count; waist circumference; blood pressure; HbA1c and lipid panel; risk of diabetes; and quality of life), compliance with and effect of the GLB-TBI and Attention Control App at 18 months.

Aim 4.1: To evaluate and integrate deep phenotype profiling (e.g. proteomics, metabolomics) and correlate findings with rehabilitation therapy and outcomes in patients with TBI.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 64 years of age
* At least 6 months post-TBI
* Moderate to severe TBI at time of injury
* BMI greater than or equal to 25
* Physician approval by week 4 of program. For those who are randomized into the attention control support group, physician approval will not be needed because information regarding physical activity and promotion will not be provided.
* Have or willing to use a smartphone or tablet

Exclusion Criteria:

* Conditions in which physical activity is contraindicated
* Not fluent in the English language
* Low cognitive function
* Residing in a hospital, acute rehabilitation setting, or skilled nursing facility
* Currently taking medication for type 2 diabetes
* Pre-existing diagnosis of an eating disorder
* Pregnancy
* Previous participants

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in weight | Baseline, 3 months, 6, months, 12 months, and 18 months
  Weight will be obtained using the same scale over the study period that is accessible to people with and without a mobility device (e.g. walker; wheelchair)

SECONDARY OUTCOMES:
Step Count | 3 months, 6 months, 12 months, and 18 months
  The Garmin Vivofit will be worn for the study duration to measure physical activity data.
Waist and Arm Circumference | Baseline, 3 months, 6 months, 12 months, and 18 months
  Waist circumference will be measured at the umbilicus and mild-upper arm circumference following American College of Sports Medicine guidelines.
Blood Pressure | Baseline, 3 months, 6 months, 12 months, and 18 months
  Using an automatic cuff (average of three readings, patient seated) diastolic and systolic scores will be recorded.
HbA1c and Lipid Panel | Baseline, 3 months, 6 months, 12 months, and 18 months
  Fasting venous sample will be obtained for blood glucose, HDL/LDL, cholesterol, and triglyceride level.
Risk of Diabetes | Baseline, 3 months, 6 months, 12 months, and 18 months
  The Framingham Heart Study diabetes risk score will be calculated using predictors including age, gender, fasting glucose, body mass index, HDL cholesterol and triglyceride levels, blood pressure, and parental history. Risk score calculator and regression model are free and used in GLB weight-loss trials. Each risk predictor is assigned points ranging from. Risk factors are combined and a total score is calculated, with higher scores designating greater 8-year risk.. The age range for this score is 45 years or older, and therefore only individuals over this age will have calculated scores. Furthermore, the minimum cut-off score is 3.
Satisfaction with Life | Baseline, 3 months, 6 months, 12 months, and 18 months
  Satisfaction with life will be measured using the Satisfaction with Life Scale (SWLS). The SWLS is a 5-item scale designed to measure global cognitive judgements of one's life satisfaction. Participants indicate how much they agree or disagree with each of the 5 items using a 7-point scale that ranges from 7-strongly agree to 1-strongly disagree. Scores are added together and a total score is calculated, with higher scores signifying higher satisfaction with life and lower scores signifying lower satisfaction with life.
Biomarkers | Baseline, 3 months, 6 months, 12 months, and 18 months
  TSH, Cortisol, IL-6, THNF, BDNF, IGF, and VEGF will be collected.
10 Meter Walk Test (10MWT) | Baseline, 3 months, 6 months, and 12 months
  Assesses walking speed in (m/s) which is correlated to mobility in the community, capacity to perform ADLs, risk of falls, re-hospitalization, and risk of cognitive decline.
6 Minute Walk Test (6MWT) | Baseline, 3 months, 6 months, and 12 months
  Assesses distance walked (rolled for wheelchair users) over 6 minutes as a sub-maximal test of aerobic capacity.
Social Support assessed by the Social Support for Diet and Exercise Behaviors Scale | Baseline, 3 months, 6 months, 12 months, and 18 months
  Social Support for Diet and Exercise Behaviors Scale is a 23-item survey including four subscales: support for healthy eating (5 items); support for physical activity (11 items); social undermining for healthy eating (5 items) and physical activity (2 items). Each item is rated on a scale of 1 to 5 (1 none; 5 very often), with respondents asked to rate support from family, friends, and coworkers. Higher scores represent greater support and internal consistency ranged from Cronbach's α 0.72-0.76.
App Feasibility and Usability using the Feasibility and Usability Survey | 6 months, 12 months, and 18 months
  The Feasibility and Usability survey includes 14 items that assesses the participant's subjective experience with the App, level of difficulty, prompting sequence, length, and understanding. Scores above 3 on the scale (1 [totally disagree] - 5 [totally agree]) indicate that the App was easy to use.
Neighborhood Walkability assessed by the Neighborhood Environment Walkability Scale (NEWS) | Baseline and 12 months
  NEWS assesses residents' perception of neighborhood design features, categorized into subscales related to physical activity, including residential density, land use mix (including both indices of proximity and accessibility), street connectivity, infrastructure for walking/cycling, neighborhood aesthetics, traffic and crime safety, and neighborhood satisfaction. Subscales are scored as a mean of items. Higher scores denote higher walkability.
Self-Reported Activities of Health using the Self-Reported Activities of Health for Health Promotion Scale | Baseline, 12 months, and 18 months
  Measure includes 28 items that assess health practices among people with disabilities and yields a total Health Practices score plus 4 subscales scores regarding Exercise, Nutrition, Health Practices, and Psychological Well Being. Items are rated on a 5-point scale from 0 'not at all' to 4 'completely.' Scores range from 0-28 with higher scores indicating higher exercise self-efficacy.
Stressful Life Events assessed by the Holmes and Rahe Stress Inventory | Baseline, 3 months, 6 months, 12 months, and 18 months
  This inventory consists of 40 life events and asks the participant to recall if any of the events happened within the previous year (e.g., death of spouse; personal illness; change in sleep). Endorsement of these events are totaled and higher scores indicate a greater amount of stressful life events. Point values for the Holmes and Rahe Stress Inventory were weighted and summed for each individual based on scoring instructions. Individuals who scored 150 points or less were categorized as low susceptibility to a health breakdown in the next two years, 151-300 points were 50% chance of health breakdown, and 301 points or more were 80% chance of health breakdown.
App Data | 6 months, 12 months, and 18 months
  The GLB TBI/Attention Control groups will both use this app. Usage and engagement will be collected.
Executive Function assessed by the Montreal Cognitive Assessment | Baseline, 3 months, and 12 months
  The MOCA is a brief, 8-section assessment of various cognitive domains including executive function, memory, language, attention, concentration, orientation, and working memory in neurologic populations. Each item on the MOCA is allocated a set of points adding up to 30.
Self-reported perceptions of habit strength assessed by the Self-Report Habit Index (SRHI) | Baseline, 3 months, and 12 months
  Self-Report Habit Index measures self-reported perceptions of habit strength for an identified behavior. The measure has high internal reliability across four studies. The measure consists of 12 items using a 7-point Likert scale ranging from "completely disagree" to "completely agree", with higher scores representing greater perception of habit strength.
Depression assessed using the Patient Health Questionnaire-8 item | Baseline, 12 months, and 18 months
  The PHQ-8 is a brief self-report measure of major depressive disorder, derived from the PHQ-9 by removing the last question regarding suicide assessment.It is considered to be a valid measure of depression for population-based studies and clinical populations, and has been used in studies of patients with physical injury. Frequency of symptoms during the last 2 weeks is assessed on a 0 (not at all) to 3 (nearly every day) scale. A cut-off score of 10 or greater is considered diagnostic for current depression
Walk Score | Baseline and 12 months
  Walk Score is publically available and measures walkability of any address using a patented system. Fore each address, Walk Score analyzes hundreds of walking routes to nearby amenities and awards points based on distance to each amenities. Scores are given on a scale of 0 to 100.
Behavioral Assessment | Baseline and 6 months
  The BAST is a 47 item, theoretically grounded, validated survey of behavioral and emotional symptoms for community-based adults with TBI. This assessment is a shortened version of the validated 77-item survey, with questions related to environmental stressors and mood removed due to repetitiveness to other questions in survey packet. Responses are asked over the past two weeks using an ordinal scale from 0 "rarely" to 5 "very often." There are 6 subscales: Negative Affect, Substance Use, Executive Function, Fatigue, Impulsivity, and Maladaptive Coping. Higher scores indicate more symptoms in those domains. This measure will be used to characterize behavioral/emotional symptoms and to explore whether these are factors that influence
General Self Efficacy | Baseline, 12 months, and 18 months
  The ten items from the General Self-Efficacy Scale (GSE) are deigned to examine goal-setting, effort investment, persistence in face of barriers and recovery from setbacks as constructs of perceived self-efficacy. The total score is the sum ranging from 10-40 and the instrument has been normed against the U.S. Adult population with a mean score of 29.48.
Behavioral Risk Factor Surveillance | Baseline, 3, 6, 12, and 18 months.
  The BRFSS is a state-based system of health surveys that collects information on health risk behaviors, preventative health practices, and health care access primarily related to chronic disease and injury. The GLB-TBI uses the two subscales of Healthy Eating and Physical Activity from the 2017 version of the BRFSS. It consists of 14 items.
MedGem | Baseline
  This is an FDA cleared and validated indirect calorimetry device. It is handheld and measures oxygen consumption (V02) to determine resting metabolic rate (RMR)
Metabolic Score Calculator (MetS) | Baseline, 3, 6, 12, and 18 months
  The metabolic score calculator will be used at all time points to determine the risk for metabolic syndrome. The following variables will be used to determine metabolic risk using the free metabolic risk calculator: gender, race and ethnicity, systolic blood pressure, fasting glucose, triglycerides, high-density lipoprotein (HDL), weight, height, and waist circumference. Scores are calculated are standardized to the general population.
Substance Use | Baseline, 12 months
  Information on substance use will be collected using the AUDIT-C (for alcohol use) and three questions regarding tobacco and non-prescriptive drug use.
CRISIS (CoRonavIruS Health Impact Survey) V0.3 Adult Baseline Form | Up to 12 months
  This self-report survey was developed by the National Institute of Mental Health. The full survey consists of 64 questions with an open-ended section at the end to elicit concerns and feedback related to the effects of COVID-19. For this current study, however, only sections on Exposure Status (10 items), Life Changes (15 items), and Emotions/Worries (7 items), and the open-ended question will be asked. Questions are asked "over the past two weeks."
PROMIS Social Isolation Short Form 4a | Up to 12 months
  The Social Isolation Short-Form 4a is taken from the Patient-Reported Outcomes Measurement Information System (PROMIS). This form assesses the perceptions of being "avoided, excluded, detached, disconnected from, or unknown by, others. There is no timeframe for the form. The measure is normed to the US population.
Media Questionnaire | Up to 12 months
  To assess media exposure and fear of media exposure during COVID-19 we have added 6 questions. These are asked "over the past two weeks." These questions address time spent watching the television, listening to radio, reading the newspaper, and searching the internet and social media. In addition, a 6th question related to fear is asked using a 5-point Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Driver, PhD, Principal Investigator — Baylor Scott & White Institute for Rehabilitation
Locations (1):
- Baylor Scott & White Institute for Rehabilitation, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Driver S, Juengst S, Reynolds M, McShan E, Kew CL, Vega M, Bell K, Dubiel R. Healthy lifestyle after traumatic brain injury: a brief narrative. Brain Inj. 2019;33(10):1299-1307. doi: 10.1080/02699052.2019.1641623. Epub 2019 Jul 12. PMID 31296066
- [Background] Driver S, Juengst S, McShan EE, Bennett M, Bell K, Dubiel R. A randomized controlled trial protocol for people with traumatic brain injury enrolled in a healthy lifestyle program (GLB-TBI). Contemp Clin Trials Commun. 2019 Jan 31;14:100328. doi: 10.1016/j.conctc.2019.100328. eCollection 2019 Jun. PMID 30775611
- [Background] Douglas M, Driver S, Callender L, Woolsey A. Evaluation of a 12-month lifestyle intervention by individuals with traumatic brain injury. Rehabil Psychol. 2019 Feb;64(1):25-36. doi: 10.1037/rep0000253. Epub 2018 Dec 20. PMID 30570330
- [Background] Reynolds M, Driver S, Bennett M. The social network - using social media to support individuals with traumatic brain injury participating in a pilot study weight-loss program. Brain Inj. 2018;32(12):1450-1454. doi: 10.1080/02699052.2018.1496480. Epub 2018 Jul 12. PMID 30325274
- [Background] Driver S, Reynolds M, Woolsey A, Callender L, Prajapati PK, Bennett M, Kramer K. Impact of a Community-Based Healthy Lifestyle Program on Individuals With Traumatic Brain Injury. J Head Trauma Rehabil. 2018 Nov/Dec;33(6):E49-E58. doi: 10.1097/HTR.0000000000000372. PMID 29385008
- [Background] Driver S, Reynolds M, Kramer K. Modifying an evidence-based lifestyle programme for individuals with traumatic brain injury. Brain Inj. 2017;31(12):1612-1616. doi: 10.1080/02699052.2017.1346286. Epub 2017 Jul 27. PMID 28750178
- [Background] Driver S, Reynolds M, Douglas M, Bennett M. Describing Weight Loss Attempts and Physical Activity Among Individuals With TBI Prior to Participation in a Weight-Loss Program. J Head Trauma Rehabil. 2018 Jan/Feb;33(1):E36-E43. doi: 10.1097/HTR.0000000000000327. PMID 28520676
- [Derived] McShan EE, Juengst S, Douglas ME, Noorbakhsh D, Calhoun S, Bennett M, Suhalka A, Dubiel R, Driver S. Efficacy of a group-based education intervention for people with traumatic brain injury: supplementary results from a 12-month randomized controlled trial. Brain Inj. 2023 Aug 24;37(10):1205-1214. doi: 10.1080/02699052.2023.2225874. Epub 2023 Jun 24. PMID 37355803
- [Derived] Juengst SB, McShan E, Conley M, Luu I, Driver S. Feasibility and Pilot Testing of Mobile Health Apps to Supplement 2 Healthy Lifestyle Interventions in Chronic Traumatic Brain Injury. J Head Trauma Rehabil. 2022 May-Jun 01;37(3):162-170. doi: 10.1097/HTR.0000000000000769. Epub 2022 Mar 15. PMID 35293364